CLINICAL TRIAL: NCT03019185
Title: A Phase 2/3 Trial of the Efficacy and Safety of Bardoxolone Methyl in Patients With Alport Syndrome
Brief Title: A Phase 2/3 Trial of the Efficacy and Safety of Bardoxolone Methyl in Patients With Alport Syndrome - CARDINAL
Acronym: CARDINAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RTA 402-C-1603
Record Dates: First submitted 2017-01-06; First posted 2017-01-12 (Estimated); Results first posted 2023-10-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Alport Syndrome
Keywords: Alport Syndrome; Bardoxolone methyl; CDDO-ME; RTA 402
MeSH Terms: conditions — Nephritis, Hereditary | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase 2 Bardoxolone Methyl (Experimental): Patients in the Phase 2 cohort will receive bardoxolone methyl throughout the study. Patients with baseline ACR ≤ 300 mg/g will be titrated to a maximum dose of 20 mg, and patients with baseline ACR > 300 mg/g will be titrated to a maximum dose of 30 mg. Adult patients (≥ 18 years of age) receiving bardoxolone methyl will start with once-daily dosing at 5 mg and will dose-escalate to 10 mg at Week 2, to 20 mg at Week 4, and then to 30 mg at Week 6 (only if baseline ACR >300 mg/g) unless contraindicated clinically and approved by the medical monitor. Patients under the age of 18 receiving bardoxolone methyl will start 5 mg every other day during the first week and begin once-daily dosing with 5 mg during the second week of the study, and then continue with once-daily dosing following the same aforementioned dose titration scheme based on baseline ACR at Weeks 2, 4, and 6.
  Interventions: Drug: Bardoxolone Methyl
- Phase 3 Bardoxolone Methyl (Active Comparator): Patients with baseline ACR ≤ 300 mg/g will be titrated to a maximum dose of 20 mg, and patients with baseline ACR > 300 mg/g will be titrated to a maximum dose of 30 mg. Adult patients (≥ 18 years of age) receiving bardoxolone methyl will start with once-daily dosing at 5 mg and will dose-escalate to 10 mg at Week 2, to 20 mg at Week 4, and then to 30 mg at Week 6 (only if baseline ACR >300 mg/g) unless contraindicated clinically and approved by the medical monitor. Patients under the age of 18 receiving bardoxolone methyl will start 5 mg every other day during the first week and begin once-daily dosing with 5 mg during the second week of the study, and then continue with once-daily dosing following the same aforementioned dose titration scheme based on baseline ACR at Weeks 2, 4, and 6.
  Interventions: Drug: Bardoxolone Methyl
- Phase 3 Placebo (Placebo Comparator): Patients randomized to placebo will remain on placebo throughout the study, undergoing sham titration.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Placebo Oral Capsule — Capsule containing an inert placebo
  Arms: Phase 3 Placebo
Drug: Bardoxolone Methyl — Bardoxolone methyl dose escalated from 5 mg to a maximum of 20 or 30 mg, depending on baseline proteinuria status.
  Other Names: RTA 402
  Arms: Phase 2 Bardoxolone Methyl; Phase 3 Bardoxolone Methyl

SUMMARY:
This international, multi-center, Phase 2/3 trial will study the safety, tolerability, and efficacy of bardoxolone methyl in qualified patients with Alport syndrome. The Phase 2 portion of the trial will be open-label and enroll up to 30 patients. The Phase 3 portion of the trial will be double-blind, randomized, placebo-controlled and will enroll up to 180 patients.

DETAILED DESCRIPTION:
This international, multi-center, Phase 2/3 trial will study the safety, tolerability, and efficacy of bardoxolone methyl in qualified patients with Alport syndrome. The Phase 2 portion of the trial will be open-label and enroll up to 30 patients. The Phase 3 portion of the trial will be double-blind, randomized, placebo-controlled and will enroll up to 180 patients.

Patients in the Phase 2 cohort will receive bardoxolone methyl throughout the study. Patients in the Phase 3 cohort will be randomized 1:1 to either bardoxolone methyl or placebo and randomization will be stratified by baseline albumin to creatinine ratio (ACR). Patients randomized to placebo will remain on placebo throughout the study, undergoing sham titration.

All patients in the study will follow the same visit and assessment schedule. Following randomization on Day 1, patients will be scheduled to be assessed during treatment at Weeks 1, 2, 4, 6, 8, 12, 24, 36, 48, 52, 64, 76, 88, 100, and 104 and by telephone contact on Days 3, 10, 21, 31, 38, and 45. Patients will not receive study drug during a 4-week withdrawal period between Weeks 48 and 52. They will re-start treatment at Week 52 at the same dose they received at Week 48 and will continue study drug treatment through Week 100. Patients will also be scheduled to be assessed at an in person follow up visit at Week 104, four weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 12 ≤ age ≤ 60 upon study consent;
* Diagnosis of Alport syndrome by genetic testing (documented mutation in a gene associated with Alport syndrome, including COL4A3, COL4A4, or COL4A5) or histologic assessment using electron microscopy;
* Screening eGFR ≥ 30 and ≤ 90 mL/min/1.73 m2. The two eGFR values collected at Screen A and Screen B visits used to determine eligibility must have a percent difference ≤ 25%;
* Albumin to creatinine ratio (ACR) ≤ 3500 mg/g at Screen B visit;
* If receiving an angiotensin-converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB), the medications must remain the same for at least 6 weeks prior to the Screen A visit and during Screening. The dosage of ACE inhibitor and/or ARB must also be stable for 2 weeks prior to the Screen A visit and remain the same through Day 1 (i.e., no change in dosage or medication). Patients not taking an ACE inhibitor and/or ARB because of a medical contraindication must have discontinued treatment at least 8 weeks prior to the Screen A visit;
* Adequate bone marrow reserve and organ function at the Screen A visit
* Able to swallow capsules;
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures;

Exclusion Criteria:

* Prior exposure to bardoxolone methyl;
* Ongoing chronic hemodialysis or peritoneal dialysis therapy;
* Renal transplant recipient;
* B-type natriuretic peptide (BNP) level > 200 pg/mL at Screen A visit;
* Uncontrolled diabetes (HbA1c > 11.0%) at Screen A visit;
* Acute dialysis or acute kidney injury within 12 weeks prior to Screen A visit or during Screening;
* Serum albumin < 3 g/dL at Screen A visit;
* History of clinically significant left-sided heart disease and/or clinically significant cardiac disease, including but not limited to any of the following:
* Uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure (BP) > 160 mm Hg or sitting diastolic BP > 100 mm Hg at Screen A visit after a period of rest;
* Systolic BP < 90 mm Hg at Screen A visit after a period of rest;
* History of malignancy within 5 years prior to Screen A visit, with the exception of localized skin or cervical carcinomas;
* Systemic immunosuppression for more than 2 weeks, cumulatively, within the 12 weeks prior to randomization or anticipated need for immunosuppression during the study;
* Untreated or uncontrolled active bacterial, fungal, or viral infection;
* Participation in other interventional clinical studies within 30 days prior to Day 1;
* Unwilling to practice acceptable methods of birth control (both males who have partners of child-bearing potential and females of childbearing potential) during Screening, while taking study drug, and for at least 30 days after the last dose of study drug is ingested;
* Women who are pregnant or breastfeeding;
* Known hypersensitivity to any component of the study drug

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 187 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (38):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Kidney Disease and Hypertension Research Services, PLLC, Phoenix, Arizona
  - Scripps Clinic, Nephrology, La Jolla, California
  - Academic Medical Research Institute, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - General Clinical Research Center - Parnassus, San Francisco, California
  - University of California San Francisco - Children's Renal Center, San Francisco, California
  - Denver Nephrologists PC, Denver, Colorado
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Emory University School of Medicine and Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boise Kidney & Hypertension Institute, Caldwell, Idaho
  - Boise Kidney & Hypertension Institute, Meridian, Idaho
  - NorthShore University Health System, Evanston, Illinois
  - Biolab Research, LLC, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota - Division of Pediatric Nephrology, Minneapolis, Minnesota
  - Children's Research Institute - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack Meridian School of Medicine, Hackensack, New Jersey
  - Nephrology Associates, PC, Flushing, New York
  - Columbia University Nephrology, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Brookview Hills Research Associates, PLLC, Winston-Salem, North Carolina
  - Akron Nephrology Associates, Akron, Ohio
  - Akron Children's Hospital, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine - Division of Pediatric Nephrology, Pittsburgh, Pennsylvania
  - The Warren Alpert Medical School of Brown University, Providence, Rhode Island
  - South Carolina Nephrology & Hypertension Center, Inc, Orangeburg, South Carolina
  - Renal Disease Research Institute, Dallas, Texas
  - Southwest Houston Research, Houston, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
- Australia (5):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Melbourne Renal Research Group, Melbourne
  - John Hunter Hospital, New Lambton Heights
  - Sydney Children's Hospital, Sydney
  - The Children's Hospital at Westmead, Westmead
- France (3):
  - CHU Grenoble- Grenoble France, La Tronche
  - CHU Lyon-Hopital Edouard Herriot, Lyon
  - Hopital Necker-Universite Paris Descartes, Paris
- Germany (2):
  - University of Medicine Gottingen, Göttingen
  - University Children's Hospital Heidelberg, Heidelberg
- Japan (10):
  - St Marianna University Hospital, Kawasaki
  - Kobe University Hospital, Kobe
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya
  - JCHO Cyukyo Hospital, Nagoya
  - Kitano Hospital, Osaka
  - Saga University Hospital, Saga
  - Saitama Children's Medical Center, Saitama
  - JCHO Sendai Hospital, Sendai
  - Juntendo University Hospital, Tokyo
  - Tokyo Metropolitan Children's Medical Center, Tokyo
- Puerto Rico Clinical & Translational Research Center, Rio Piedras, Puerto Rico
- Spain (3):
  - Servicio de Nefrologia pediatrica, Barcelona
  - Fundacio Puigvert, Barcelona
  - Hospital Virgen de la Arrixaca, El Palmar
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Warady BA, Pergola PE, Agarwal R, Andreoli S, Appel GB, Bangalore S, Block GA, Chapman AB, Chin MP, Gibson KL, Goldsberry A, Iijima K, Inker LA, Kashtan CE, Knebelmann B, Mariani LH, Meyer CJ, Nozu K, O'Grady M, Rheault MN, Silva AL, Stenvinkel P, Torra R, Chertow GM. Effects of Bardoxolone Methyl in Alport Syndrome. Clin J Am Soc Nephrol. 2022 Dec;17(12):1763-1774. doi: 10.2215/CJN.02400222. Epub 2022 Nov 21. PMID 36411058
- [Derived] Chertow GM, Appel GB, Andreoli S, Bangalore S, Block GA, Chapman AB, Chin MP, Gibson KL, Goldsberry A, Iijima K, Inker LA, Knebelmann B, Mariani LH, Meyer CJ, Nozu K, O'Grady M, Silva AL, Stenvinkel P, Torra R, Warady BA, Pergola PE. Study Design and Baseline Characteristics of the CARDINAL Trial: A Phase 3 Study of Bardoxolone Methyl in Patients with Alport Syndrome. Am J Nephrol. 2021;52(3):180-189. doi: 10.1159/000513777. Epub 2021 Mar 31. PMID 33789284
- [Derived] Kashtan CE, Gross O. Clinical practice recommendations for the diagnosis and management of Alport syndrome in children, adolescents, and young adults-an update for 2020. Pediatr Nephrol. 2021 Mar;36(3):711-719. doi: 10.1007/s00467-020-04819-6. Epub 2020 Nov 6. PMID 33159213
- See also: Website for the CARDINAL study — https://www.cardinalclinicaltrial.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CARDINAL Phase 2 and Phase 3 were conducted under the same protocol. Participants enrolled in Phase 2 were not allowed to enroll in Phase 3.
Groups:
- Phase 2 Bardoxolone Methyl: Participants who received bardoxolone methyl capsules at a starting dose of 5 mg and titrated up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily in the Cardinal Phase 2 Study
- Phase 3 Placebo: Participants who received placebo (with sham titration) in the Cardinal Phase 3 Study
- Phase 3 Bardoxolone Methyl: Participants who received bardoxolone methyl capsules at a starting dose of 5 mg and titrated up to a maximal dose of 20 mg (participants with UACR less than or equal to 300 mg/g) or 30 mg (participants with UACR greater than 300 mg/g) daily in the Cardinal Phase 3 Study
Period: Overall Study
Arm/Group | Phase 2 Bardoxolone Methyl | Phase 3 Placebo | Phase 3 Bardoxolone Methyl
Started | 30 | 80 | 77
Completed | 24 | 79 | 75
Not Completed | 6 | 1 | 2
Not completed — Lost to Follow-up | 3 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Inability to continue due to increased serum creatinine | 1 | 0 | 0
Not completed — ESKD Resulting in Kidney Transplant | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 2 Bardoxolone Methyl | Phase 3 Placebo | Phase 3 Bardoxolone Methyl | Total
Number analyzed (Participants) | 30 | 80 | 77 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.63 (12.557) | 39.6 (16.03) | 38.8 (14.55) | 39.9 (14.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 48 | 43 | 109
  Male | 12 | 32 | 34 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 10 | 9 | 22
  Not Hispanic or Latino | 27 | 70 | 68 | 165
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 12 | 14 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 2 | 3 | 8
  White | 26 | 63 | 55 | 144
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 30 | 57 | 54 | 141
  Japan | 0 | 9 | 12 | 21
  Australia | 0 | 1 | 4 | 5
  France | 0 | 5 | 2 | 7
  Germany | 0 | 3 | 2 | 5
  Spain | 0 | 5 | 3 | 8
Baseline estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 54.17 (24.075) | 62.63 (18.234) | 62.74 (17.719) | 61.32 (19.227)
Baseline urine albumin-to-creatinine ratio (UACR) [Geometric Mean (Full Range); unit: mg/g] | 147.83 [2.4 to 1600.0] | 134.45 [1.2 to 3031.0] | 148.09 [2.1 to 3495.0] | 142.05 [1.2 to 3495.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) After 12 Weeks of Treatment (Phase 2)
Description: To assess the change in eGFR from baseline to week 12 (Phase 2). Estimated Glomerular filtration rate (eGFR) indicates how well the kidneys are filtering waste from the blood. The higher the eGFR number, the better the kidney function.
Time Frame: Baseline through 12 weeks after participant receives the first dose in the Phase 2 study
Population: Intent-to-treat population (all enrolled patients)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Phase 2 Bardoxolone Methyl
Number analyzed (Participants) | 30
mL/min/1.73 m^2 | 13.37 (1.4111)
Statistical Analysis 1: Comparison: Phase 2 Bardoxolone Methyl; Test type: Superiority — A formal test of mean change from baseline in eGFR ≠ 0 was conducted at Week 12; p < 0.0001, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 12 were included. Missing data were not imputed; LS Mean change from baseline = 13.37, 95% CI 2-sided [10.48 to 16.27], Standard Error of Mean 1.4111

2. Primary Outcome: Change From Baseline in eGFR After 48 Weeks of Treatment (Phase 3)
Description: To assess the change in eGFR from baseline to week 48 (Phase 3). Estimated Glomerular filtration rate (eGFR) indicates how well the kidneys are filtering waste from the blood. The higher the eGFR number, the better the kidney function.
Time Frame: Baseline through 48 weeks after participant receives the first dose in the Phase 3 study
Population: Intent-to-treat population (all randomized patients)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Phase 3 Placebo | Phase 3 Bardoxolone Methyl
Number analyzed (Participants) | 80 | 77
mL/min/1.73 m^2 | -4.77 (1.248) | 4.71 (1.307)
Statistical Analysis 1: Comparison: Phase 3 Placebo vs Phase 3 Bardoxolone Methyl; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 48 were included. Missing data were not imputed; LS Mean difference (Net) = 9.49, 97.5% CI 2-sided [5.38 to 13.60], Standard Error of Mean 1.813 — Difference is bardoxolone methyl - placebo

3. Primary Outcome: Change From Baseline in eGFR After 100 Weeks of Treatment (Phase 3)
Description: To assess the change in eGFR from baseline to week 100 (Phase 3). Estimated Glomerular filtration rate (eGFR) indicates how well the kidneys are filtering waste from the blood. The higher the eGFR number, the better the kidney function.
Time Frame: Baseline through 100 weeks after participant receives the first dose in the Phase 3 study
Population: Intent-to-treat population (all randomized patients)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Phase 3 Placebo | Phase 3 Bardoxolone Methyl
Number analyzed (Participants) | 80 | 77
mL/min/1.73 m^2 | -8.45 (1.478) | -0.81 (1.556)
Statistical Analysis 1: Comparison: Phase 3 Placebo vs Phase 3 Bardoxolone Methyl; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 100 (excluding Week 52) were included. Missing data were not imputed; LS Mean difference (Net) = 7.65, 95% CI 2-sided [3.41 to 11.89], Standard Error of Mean 2.144 — Difference is bardoxolone methyl - placebo

4. Secondary Outcome: Change From Baseline in eGFR After 48 Weeks of Treatment (Phase 2)
Description: To assess the change from baseline in eGFR in bardoxolone methyl-treated patients at Week 48. Estimated Glomerular filtration rate (eGFR) indicates how well the kidneys are filtering waste from the blood. The higher the eGFR number, the better the kidney function.
Time Frame: Baseline through 48 weeks after participant receives the first dose in the Phase 2 study
Population: Intent-to-treat population (all enrolled patients)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Phase 2 Bardoxolone Methyl
Number analyzed (Participants) | 30
mL/min/1.73 m^2 | 7.4 (1.9451)
Statistical Analysis 1: Comparison: Phase 2 Bardoxolone Methyl; Test type: Superiority — A formal test of mean change from baseline in eGFR ≠ 0 was conducted at Week 48; p = 0.0008, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 48 were included. Missing data were not imputed; LS Mean change from baseline = 7.40, 95% CI 2-sided [3.40 to 11.39], Standard Error of Mean 1.9451

5. Secondary Outcome: Change From Baseline in eGFR After 100 Weeks of Treatment (Phase 2)
Description: To assess the change from baseline in eGFR in bardoxolone methyl-treated patients at Week 100. Estimated Glomerular filtration rate (eGFR) indicates how well the kidneys are filtering waste from the blood. The higher the eGFR number, the better the kidney function.
Time Frame: Baseline through 100 weeks after participant receives the first dose in the Phase 2 study
Population: Intent-to-treat population (all enrolled patients)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Phase 2 Bardoxolone Methyl
Number analyzed (Participants) | 30
mL/min/1.73 m^2 | 4.28 (1.7484)
Statistical Analysis 1: Comparison: Phase 2 Bardoxolone Methyl; Test type: Superiority — A formal test of mean change from baseline in eGFR ≠ 0 was conducted at Week 100; p = 0.0150, Mixed Models Analysis; Available data from analysis visits Week 1 to Week 100 (excluding Week 52) were included. Missing data were not imputed; LS Mean change from baseline = 4.28, 95% CI 2-sided [0.84 to 7.72], Standard Error of Mean 1.7484

6. Secondary Outcome: Change From Baseline in eGFR at Week 52 Following a 4-week Drug Treatment Withdrawal Period (Phase 3)
Description: To assess the change in eGFR from baseline to week 52 following a 4-week drug treatment withdrawal period (Phase 3). Estimated Glomerular filtration rate (eGFR) indicates how well the kidneys are filtering waste from the blood. The higher the eGFR number, the better the kidney function.
Time Frame: Baseline through 52 weeks after participant receives the first dose in the Phase 3 study (or 4 weeks after last dose for patients who discontinued early in the first year)
Population: Intent-to-treat population (all randomized patients)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Phase 3 Placebo | Phase 3 Bardoxolone Methyl
Number analyzed (Participants) | 80 | 77
mL/min/1.73 m^2 | -6.08 (1.243) | -0.99 (1.253)
Statistical Analysis 1: Comparison: Phase 3 Placebo vs Phase 3 Bardoxolone Methyl; Test type: Superiority; p = 0.0021, ANCOVA; Missing eGFR data were imputed using multiple imputation based on the treatment group to which the patient was assigned; LS Mean difference (Net) = 5.09, 97.5% CI 2-sided [1.37 to 8.80], Standard Error of Mean 1.656 — Difference is bardoxolone methyl - placebo

7. Secondary Outcome: Change From Baseline in eGFR at Week 104 Following a 4-week Drug Treatment Withdrawal Period (Phase 3)
Description: To assess the change in eGFR from baseline to week 104 following a 4-week drug treatment withdrawal period (Phase 3). Estimated Glomerular filtration rate (eGFR) indicates how well the kidneys are filtering waste from the blood. The higher the eGFR number, the better the kidney function.
Time Frame: Baseline through 104 weeks after participant receives the first dose in the Phase 3 study (or 4 weeks after last dose for patients who discontinued early in the second year)
Population: Intent-to-treat population (all randomized patients)
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Phase 3 Placebo | Phase 3 Bardoxolone Methyl
Number analyzed (Participants) | 80 | 77
mL/min/1.73 m^2 | -8.84 (1.353) | -4.52 (1.395)
Statistical Analysis 1: Comparison: Phase 3 Placebo vs Phase 3 Bardoxolone Methyl; Test type: Superiority; p = 0.0232, ANCOVA; Missing eGFR data were imputed using multiple imputation based on the treatment group to which the patient was assigned; LS Mean difference (Net) = 4.26, 95% CI 2-sided [0.58 to 7.94], Standard Error of Mean 1.876 — Difference is bardoxolone methyl - placebo

ADVERSE EVENTS:
Time Frame: 104 weeks
Arm/Group | Phase 2 Bardoxolone Methyl | Phase 3 Placebo | Phase 3 Bardoxolone Methyl
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/80 | 0/77
Serious Adverse Events (participants affected / at risk) | 6/30 | 15/80 | 8/77
Other Adverse Events (participants affected / at risk) | 29/30 | 76/80 | 75/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 Bardoxolone Methyl (N=30) | Phase 3 Placebo (N=80) | Phase 3 Bardoxolone Methyl (N=77)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Status migrainosus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 3 (3) | 2 (2) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 Bardoxolone Methyl (N=30) | Phase 3 Placebo (N=80) | Phase 3 Bardoxolone Methyl (N=77)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 2 (4)
Deafness (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 2 (2)
Hyperparathyroidism secondary (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 13 (16) | 8 (9)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (4) | 7 (7)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 6 (7) | 12 (14)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (7)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (10) | 11 (15) | 13 (19)
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 3 (5) | 3 (4) | 7 (9)
Asthenia (General disorders) | 0 (0) | 3 (3) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 6 (7) | 12 (16) | 14 (18)
Malaise (General disorders) | 3 (3) | 0 (0) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 6 (6)
Oedema peripheral (General disorders) | 7 (8) | 10 (15) | 12 (18)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Ear infection (Infections and infestations) | 1 (1) | 1 (2) | 2 (2)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 7 (7) | 6 (6)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 24 (29) | 18 (27)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (2) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 2 (3) | 7 (8) | 6 (7)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 8 (10) | 12 (15)
Urinary tract infection (Infections and infestations) | 2 (5) | 5 (9) | 3 (8)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 4 (5)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (17) | 2 (2) | 36 (41)
Albumin urine present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 1 (1) | 19 (22)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 9 (11) | 5 (7)
Blood creatinine increased (Investigations) | 1 (1) | 8 (8) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 2 (2) | 4 (4)
Brain natriuretic peptide abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 3 (4) | 3 (3) | 11 (23)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1) | 4 (4)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 2 (2) | 5 (5)
Urine albumin/creatinine ratio increased (Investigations) | 2 (2) | 7 (8) | 8 (9)
Vitamin D decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 10 (12)
Weight increased (Investigations) | 0 (0) | 6 (7) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 3 (3) | 6 (8) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (12) | 5 (9) | 11 (19)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 13 (16) | 9 (9)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 (43) | 27 (45) | 38 (72)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (6) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 7 (8)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 12 (13) | 3 (3)
Dysgeusia (Nervous system disorders) | 4 (4) | 1 (1) | 4 (5)
Headache (Nervous system disorders) | 6 (9) | 16 (31) | 16 (28)
Migraine (Nervous system disorders) | 2 (2) | 2 (3) | 1 (4)
Migraine without aura (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Periodic limb movement disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Albuminuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (5) | 6 (6) | 7 (7)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4) | 8 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 7 (14)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 4 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (8) | 8 (9) | 7 (7)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (8):
  • Study Protocol: US Protocol (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03019185/Prot_000.pdf
  • Study Protocol: US Protocol Addendum (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03019185/Prot_001.pdf
  • Study Protocol: Europe Protocol (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03019185/Prot_002.pdf
  • Study Protocol: Germany Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03019185/Prot_003.pdf
  • Study Protocol: France Spain UK Protocol (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03019185/Prot_004.pdf
  • Study Protocol: France Spain UK Protocol Addendum (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03019185/Prot_005.pdf
  • Statistical Analysis Plan: Phase 2 SAP (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03019185/SAP_006.pdf
  • Statistical Analysis Plan: Phase 3 SAP (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT03019185/SAP_007.pdf